CLINICAL TRIAL: NCT04492163
Title: EF-33: An Open-Label Pilot Study of OPTUNE® (TTFields, 200 Khz) With High Density Transducer Arrays for the Treatment of Recurrent Glioblastoma
Brief Title: Open-Label Pilot Study of OPTUNE® With High Density Transducer Arrays for the Treatment of Recurrent GBM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovoCure GmbH (Industry)
Responsible Party: Sponsor
Organization: NovoCure Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF-33
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; Recurrent Glioblastoma; GBM; Treatment; Minimal Toxicity; TTFields; Tumor Treating Fields; NovoCure
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Single group assignment
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: TTFields (Experimental): Patients receive continuous TTFields treatment using the Optune® System with high intensity transducer arrays.
  Interventions: Device: TTFields

INTERVENTIONS:
Device: TTFields — TTFields treatment will consist of wearing four electrically insulated electrode arrays on the head. The treatment enables the patient to maintain regular daily routine.
  Other Names:
  • TTFields

SUMMARY:
This is a prospective, open-label, single arm, historical control pilot study aimed to test the effectiveness and safety of TTFields delivered through high intensity arrays in recurrent glioblastoma.

The Optune® System is an investigational , portable, battery operated medical device in this study delivering 200 kHz TTFields to the brain using high intensity transducer arrays for the treatment of patients at the age of 18 years or older with first or second recurrence of Glioblastoma Multiforme (GBM)

DETAILED DESCRIPTION:
Optune® is a medical device that has been approved for the treatment of recurrent and newly diagnosed glioblastoma (GBM) by the Food and Drug Administration (FDA) in the United States. Optune® has obtained a CE mark in Europe for recurrent and newly diagnosed GBM.

TTFields intensity has been shown to be positively correlated with patient outcome. The new transducer array design is expected to reduce skin heating and thus enable delivery of higher TTFields intensities while keeping the safety profile of the treatment unchanged.

The purpose of the study is to test if delivering TTFields using high intensity transducer arrays for recurrent GBM significantly improves the clinical outcome of patients, compared to using the standard transducer arrays.

The study will enroll 25 patients.

All patients included in this clinical investigation are patients with histologically confirmed diagnosis of GBM with first or second radiological disease progression per RANO criteria.

In addition, all patients must meet all eligibility criteria.

Baseline assessments will be performed to confirm patient eligibility in the study.

Enrolled patients will be treated continuously with the device until disease progression per RANO criteria or 18 months (the earlier of the two) unless any of the treatment discontinuation conditions described under criteria for patient withdrawal or termination are met.

Concurrent brain directed antitumor therapy or procedures beyond TTFields is prohibited.

TTFields treatment will start within 28 days following signing the informed consent.

After the initial visit, subjects will continue treatment at home, while pursuing normal daily routines. Subjects are required to use the device for at least 18 hours a day. Short breaks in treatment for personal hygiene and other personal needs is allowed. Total usage time will be recorded and provided to the sponsor.

Subjects will be required to return to the clinic every 4 weeks and every 8 weeks after first 12 visits, until disease progression. At each study visit an examination by a physician and a routine laboratory examination will be performed.

A contrast enhanced MRI of the head will be performed at baseline and every 4 weeks for the first 24 weeks and then at least every 12 weeks, until disease progression.

A post-treatment termination visit will be performed approximately 30 days after discontinuation of TTfields treatment or disease progression (the latter of the two).

Following disease progression, subjects will be contacted once per month by telephone to answer basic questions about their health status.

Pathological analysis of GBM tumor samples, which may be obtained prior and during the study period, will be performed based on subjects' consent to have an experimental pathological examination of their tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of GBM according to WHO classification criteria.
2. Age ≥ 18 years
3. Not a candidate for further radiotherapy or additional resection of residual tumor.
4. Patients with first or second radiological disease progression per RANO criteria documented by MRI within 4 weeks prior to starting therapy with the following restriction: disease progression must be either growth of the enhancing lesion or a new lesion.
5. Karnofsky performance status ≥ 70
6. Life expectancy ≥ least 3 months
7. Participants of childbearing age must use highly effective contraception. An effective method of birth control is defined as one that results in a failure rate of less than 1% per year when used consistently and correctly. The Investigator must approve the selected method, and may consult with a gynecologist as needed.
8. All patients must understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
9. Treatment start date at least 4 weeks out from brain surgery chemotherapy or irradiation therapy.

Exclusion Criteria:

1. Infratentorial or leptomeningeal disease
2. Treatment with Optune® (for newly diagnosed or recurrent disease) prior to enrollment.
3. Participation in another clinical treatment study during screening and treatment phase of the study.
4. Pregnancy or breast-feeding.
5. Significant co-morbidities at baseline, as determined by the investigator:

   1. Thrombocytopenia (platelet count < 100 x 103/μL)
   2. Neutropenia (absolute neutrophil count < 1 x 103/μL)
   3. CTC grade 4 non-hematological Toxicity (except for alopecia, nausea, vomiting)
   4. Significant liver function impairment - AST or ALT > 3 times the upper limit of normal
   5. Total bilirubin > 1.5 x upper limit of normal
   6. Significant renal impairment (serum creatinine > 1.7 mg/dL, or > 150 µmol/l)
   7. History of any psychiatric condition that might impair patient's ability to understand or comply with the requirements of the study or to provide consent
6. Implanted pacemaker, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
7. Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness)
8. Admitted to an institution by administrative or court order.
9. Known allergies to medical adhesives or hydrogel

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 18 Months
  PFS will be measured from the date of enrollment to date of progression (in months) based on RANO citeria.

SECONDARY OUTCOMES:
Overall Survival (OS) | 18 Months
  Survival will be measured from date of enrollment until date of death.
Progression Free Survival at 6 months (PFS6) | 18 Months
  The analysis will be estimated proportions of patients who are progression-free at 6 months based on the RANO criteria following the time of enrollment.
1-year and 2-year survival rates | 24 Months
  The analyses will be performed based on estimated proportions of patients who are alive at one and two years following enrollment.
Overall radiological response | 18 Months
  The percentage of patients who had either complete response or partial response per RANO criteria following enrollment
Severity and frequency of adverse events | 18 Months
  The analyses will be performed based on the incidence, severity, frequency of adverse events, and their association with study treatments
Pathological changes in resected GBM tumors following study treatment | 18 Months
  Pathological changes in the tumors of patients who consented to have pathological analysis of their tumors and also underwent another surgical resection while on the study
Dependence of Progression Free Survival on TTFields dose delivered to the tumor bed | 18 months
Dependence of Overall Survival on TTFields dose delivered to the tumor bed | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Josef Vymazal, MD, DSc, Principal Investigator — Nemocnice Na Homolce (Na Homolce Hospital
Locations (1):
- Nemocnice Na Homolce, Prague, Czechia

REFERENCES:
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Background] Giladi M, Schneiderman RS, Voloshin T, Porat Y, Munster M, Blat R, Sherbo S, Bomzon Z, Urman N, Itzhaki A, Cahal S, Shteingauz A, Chaudhry A, Kirson ED, Weinberg U, Palti Y. Mitotic Spindle Disruption by Alternating Electric Fields Leads to Improper Chromosome Segregation and Mitotic Catastrophe in Cancer Cells. Sci Rep. 2015 Dec 11;5:18046. doi: 10.1038/srep18046. PMID 26658786
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Pless M, Weinberg U. Tumor treating fields: concept, evidence and future. Expert Opin Investig Drugs. 2011 Aug;20(8):1099-106. doi: 10.1517/13543784.2011.583236. Epub 2011 May 9. PMID 21548832
- [Background] Mun EJ, Babiker HM, Weinberg U, Kirson ED, Von Hoff DD. Tumor-Treating Fields: A Fourth Modality in Cancer Treatment. Clin Cancer Res. 2018 Jan 15;24(2):266-275. doi: 10.1158/1078-0432.CCR-17-1117. Epub 2017 Aug 1. PMID 28765323
- [Background] Giladi M, Munster M, Schneiderman RS, Voloshin T, Porat Y, Blat R, Zielinska-Chomej K, Haag P, Bomzon Z, Kirson ED, Weinberg U, Viktorsson K, Lewensohn R, Palti Y. Tumor treating fields (TTFields) delay DNA damage repair following radiation treatment of glioma cells. Radiat Oncol. 2017 Dec 29;12(1):206. doi: 10.1186/s13014-017-0941-6. PMID 29284495
- [Background] Taphoorn MJB, Dirven L, Kanner AA, Lavy-Shahaf G, Weinberg U, Taillibert S, Toms SA, Honnorat J, Chen TC, Sroubek J, David C, Idbaih A, Easaw JC, Kim CY, Bruna J, Hottinger AF, Kew Y, Roth P, Desai R, Villano JL, Kirson ED, Ram Z, Stupp R. Influence of Treatment With Tumor-Treating Fields on Health-Related Quality of Life of Patients With Newly Diagnosed Glioblastoma: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):495-504. doi: 10.1001/jamaoncol.2017.5082. PMID 29392280
- [Background] Ballo MT, Urman N, Lavy-Shahaf G, Grewal J, Bomzon Z, Toms S. Correlation of Tumor Treating Fields Dosimetry to Survival Outcomes in Newly Diagnosed Glioblastoma: A Large-Scale Numerical Simulation-Based Analysis of Data from the Phase 3 EF-14 Randomized Trial. Int J Radiat Oncol Biol Phys. 2019 Aug 1;104(5):1106-1113. doi: 10.1016/j.ijrobp.2019.04.008. Epub 2019 Apr 23. PMID 31026557